CLINICAL TRIAL: NCT00359996
Title: Improving Diabetes Care Collaboratively in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9886 (AHRQ R01 HS10479)
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes
Keywords: diabetes; quality improvement; community health center; health disparities
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health disparities collaborative (Active Comparator): The HDC incorporates rapid quality improvement (QI), a chronic care model, and best practices. This study determines if the HDC improves diabetes care and whether more intensive interventions with additional learning sessions for health centers, provider training in behavioral change, and patient empowerment materials enhance care further.
  Interventions: Behavioral: health disparities collaborative
- Control (Active Comparator): No additional educational sessions added to usual care of patients.
  Interventions: Other: No additional educational sessions

INTERVENTIONS:
Behavioral: health disparities collaborative — The HDC incorporates rapid quality improvement (QI), a chronic care model, and best practices. This study determines if the HDC improves diabetes care and whether more intensive interventions with additional learning sessions for health centers, provider training in behavioral change, and patient empowerment materials enhance care further.
  Arms: Health disparities collaborative
Other: No additional educational sessions
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether a quality improvement intervention including rapid quality improvement, a chronic care model, and best practices improves diabetes care in community health centers and whether more intensive interventions enhance care further.

DETAILED DESCRIPTION:
In 1998 the Health Resources and Services Administration's Bureau of Primary Health Care began the Health Disparities Collaborative (HDC) to improve chronic disease management in community health centers (HC) nationwide. The HDC incorporates rapid quality improvement (QI), a chronic care model, and best practices. This study determines if the HDC improves diabetes care and whether more intensive interventions with additional learning sessions for health centers, provider training in behavioral change, and patient empowerment materials enhance care further.

ELIGIBILITY:
Inclusion Criteria:

- patients with diabetes age 18-75 years

Exclusion Criteria:

Pregnant women

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6993 (Actual)
Dates: Start 2000-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c | 4 years
  Change in hemoglobin A1c from baseline

SECONDARY OUTCOMES:
Lipid levels | 4 years
  Change in Lipid blood levels from baseline
Blood pressure | 4 years
  Change in BP from baseline
Urine microalbumin levels | 4 years
  Change in urine micralbumin levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marshall H Chin, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Chin MH, Drum ML, Guillen M, Rimington A, Levie JR, Kirchhoff AC, Quinn MT, Schaefer CT. Improving and sustaining diabetes care in community health centers with the health disparities collaboratives. Med Care. 2007 Dec;45(12):1135-43. doi: 10.1097/MLR.0b013e31812da80e. PMID 18007163